CLINICAL TRIAL: NCT03975205
Title: A Bio Equivalence Study of DOXIL and Doxorubicin in Subjects With Lymphoma, Leukemia and Carcinoma
Brief Title: To Study the Concentration Level of, Doxil, and Doxorubicin at Various Time Frames
Acronym: Doxil
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sutphin Drugs (Industry)
Collaborators: Bharath Charitable Cancer Hospital and Institute (Other)
Responsible Party: Principal Investigator, Dr. Ajai Prakash, President, Sutphin Drugs
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Global CRO Doxil
Record Dates: First submitted 2019-06-03; First posted 2019-06-05 (Actual); Last update posted 2019-06-05 (Actual); Status verified 2019-06

CONDITIONS: Lymphoma Leukemia
MeSH Terms: interventions — Doxorubicin; liposomal doxorubicin

STUDY DESIGN:
Intervention Model Description: A Phase 1, single-blind, randomized, two-way, crossover Bio-equivalence study of Intravenously administered Doxorubicin in Patients With lymphomas, leukemia's and carcinoma That Has Progressed or Recurred After Platinum-based Chemotherapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Doxil (Active Comparator): This group of patients will receive Intravenous Doxil of 50mgm/m2 over 15 minutes and plasma concentration will be measured at time Frame: 0, 1, 2, 3, 4, 8, 12, 24, 48 and 72 hours. Cycle is defined as 28 days
  Interventions: Drug: Doxorubicin
- doxorubicin (Experimental): This group of patients will receive Intravenous Doxorubicin of 50mgm/m2 over 15 minutes and plasma concentration will be measured at time Frame: 0, 1, 2, 3, 4, 8, 12, 24, 48 and 72 hours. Cycle is defined as 28 days
  Interventions: Drug: Doxorubicin

INTERVENTIONS:
Drug: Doxorubicin — To measure bioavailabity of Doxil versus Doxorubicin
  Other Names: Doxil

SUMMARY:
Doxil or Doxorubicin to be administered was administered in a dose of 50 mg/m2 as infusion over 15 minutes. Blood samples to be obtained at 0, 1, 2, 3, 4, 8, 12, 24, 48 and 72 hours

DETAILED DESCRIPTION:
Comparison of AUC in a single dose of Doxorubicin vs single dose of Doxil [ Time Frame: 0, 1, 2, 3, 4, 8, 12, 24, 48 and 72 hours. Cycle is defined as 28 days) The primary objective of this study is to determine the pharmacokinetic equivalence of Doxorubicin and Doxil as a single dose in patients with carcinomas, lymphomas and leukemia's. The outcome measure will be determined by analyzing the concentration from each patient at pre-specified time points and calculating Area under the curve (AUC) and Peak Plasma Concentration (C max)to determine % variability between doxorubicin and Doxil within each patient.

ELIGIBILITY:
Inclusion Criteria:

* Ages Eligible for Study: 18 Years to 75 Years (Adult, Older Adult) Sexes Eligible for Study: All Accepts Healthy Volunteers: No Criteria

Inclusion Criteria:

Have confirmed diagnosis of lymphomas. leukemia's and carcinoma to be treated with Doxil or Doxorubin Have a normal left ventricular ejection fraction (LVEF) based on institutional ranges.

Be >/= 18 and </= 75 years of age Sign a written Institutional Review Board (IRB)-approved informed consent form Have a negative pregnancy test, if patient is of child-bearing potential. Agree to use effective contraceptive methods during the study (nonsterile patients of childbearing potential) Have acceptable liver function, renal function and hematologic status based on the institution.

Exclusion criteria Any Medical related exclusion criteria as per the institution. Are unwilling or unable to comply with procedures required in this protocol Have known infection with human immunodeficiency virus (HIV), hepatitis B, or hepatitis C Have a serious nonmalignant disease (e.g., hydronephrosis, liver failure, significantly impaired hepatic function, or other conditions) that could compromise protocol objectives in the opinion of the investigator and/or the sponsor Are currently receiving any other investigational agent Have exhibited allergic reactions to doxorubicin or a similar structural compound

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2019-07-01 (Estimated); Primary Completion 2019-10-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Bioavailability of Doxil versus Doxorubicin | 72 hours . Cycle defined as 28 days
  Intravenous Doxil versus Doxorubicin of 50mgm/m2 over 15 minutes and plasma concentration will be measured at time Frame: 0, 1, 2, 3, 4, 8, 12, 24, 48 and 72 hours. Cycle is defined as 28 days.
  Maximum observed plasma concentration of doxorubicin versus Doxil in participants at time Frame: 0, 1, 2, 3, 4, 8, 12, 24, 48 and 72 hours. Cycle is defined as 28 days.

CONTACTS AND LOCATIONS:
Locations (1):
- Bharat Cancer Hospital, Surat, Gujarat, India

IPD SHARING:
Plan to Share IPD: No